CLINICAL TRIAL: NCT02117830
Title: A Thorough QT/QTc Study to Assess the Effects of Androxal in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Repros Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: ZA-108
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2014-06-16 (Estimated); Status verified 2014-06

CONDITIONS: Healthy
Keywords: To determine; effects; once; daily; oral doses; Androxal
MeSH Terms: interventions — Enclomiphene; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Androxal 25 mg (Experimental)
  Interventions: Drug: Androxal 25 mg capsules
- Androxal 250 mg (Experimental): supratherapeutic dose
  Interventions: Drug: Androxal 250 Capsules
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Capsules
- Moxifloxacin 400 mg (Other): positive control
  Interventions: Drug: Moxifloxacin 400 mg

INTERVENTIONS:
Drug: Androxal 25 mg capsules
  Arms: Androxal 25 mg
Drug: Androxal 250 Capsules
  Arms: Androxal 250 mg
Drug: Placebo Capsules
  Arms: Placebo
Drug: Moxifloxacin 400 mg
  Arms: Moxifloxacin 400 mg

SUMMARY:
This is a Phase I, single-site, randomized, double-blinded, double-dummy, placebo- and positive-controlled, 4-period crossover study to evaluate the effect of two dose levels of Androxal on cardiac repolarization. Baseline ECGs will be obtained prior to dosing in each Period and ECGs will be obtained during expected peak plasma concentrations of Androxal and the positive control.

In each Treatment Period subjects will be admitted to a Clinical Research Unit where study drug will be administered as three (3) daily single doses. Treatment Periods will be separated by a washout of at least 7 days between Periods.

ELIGIBILITY:
Inclusion Criteria:

1. Generally healthy males as determined by history and physical examination
2. Between the ages of 18 and 60, inclusive
3. Clinical laboratory test results within the normal reference ranges for the investigative site or results with acceptable deviations that are judged by the principal investigator to be not clinically significant
4. Vital signs (after 5 minutes resting in a supine position)

   * Systolic blood pressure (SBP) 90-140 mmHg, and
   * Diastolic blood pressure (DBP) 50-90 mmHg, and
   * Pulse 45-100 bpm Note: subjects with vital signs outside the above ranges may be eligible for the study if the Investigator feels that the results are not clinically significant and will not impact study conduct.
5. Body mass index (BMI) ≥25 to ≤42 kg/m2 at Screening
6. Are reliable and willing to be available for the duration of the study, abiding by the policies and procedures of the clinical trials unit
7. Have given written informed consent
8. Subject must be able to speak, read and understand English or Spanish and be willing and able to provide written informed consent in English or Spanish on an Institutional Review Board (IRB)-approved form prior to the initiation of any study procedures. Subject must have signed and dated a written informed consent form (ICF) before undergoing any study related activities, including discontinuation of any prohibited medications.

Exclusion Criteria:

1. Repros employee or investigative site personnel and their immediate families
2. Participation in a clinical trial within the past 30 days or receipt of any investigational agent or study treatment within 30 days or 5 half-lives, whichever is longer, prior to Screening
3. Known hypersensitivity to Clomid
4. Known allergy to moxifloxacin
5. Abnormal electrocardiogram that, after the option of repeating any such findings, in the opinion of the Investigator and/or Sponsor may interfere with any aspect of study conduct or interpretation of results including:

   * an abnormality of cardiac rhythm other than sinus arrhythmia
   * QTcF > 450 msec
   * QTcF < 300 msec
   * PR interval >200 msec
   * QRS > 110 msec
   * abnormal T wave morphology that will impair the ability to measure the QT interval reliably
6. History of congenital long QT syndrome or known history of QTc interval prolongation or family history of congenital long QT syndrome
7. Evidence of significant cardiac disease, for example, arrhythmia or unexplained syncope within the last year
8. History of myocardial infarction, unstable angina, symptomatic heart failure, ventricular dysrhythmia,
9. History of thrombophlebitis, thromboembolic disorder or cerebrovascular accident
10. Evidence of significant respiratory or hepatic disease
11. Use of cigarettes or any tobacco product within 2 weeks prior to Screening and while participating in the study
12. Use of any medications other than acetaminophen or aspirin (prescription or over-the-counter), herbal tea , energy drinks, supplements, within 5 days of dosing (prior to first dose of study medications), with the exception of those approved by the Investigator and Sponsor
13. Use of drugs of abuse and/or positive findings on drug screen
14. Known active infection with HIV or hepatitis B or C.

Ages: 18 Years to 60 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 54 (Estimated)
Dates: Start 2014-04; Primary Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
The placebo-subtracted change of the QTc interval from Baseline (ΔΔQTc) defined as: the change of QTc from the subject-specific and period-specific Baseline (ΔQTc), less the time-matched placebo value of change of QTc | 64 days
  The placebo-subtracted change of the QTc interval from Baseline (ΔΔQTc) defined as: the change of QTc from the subject-specific and period-specific Baseline (ΔQTc), less the time-matched placebo value of change of QTc